CLINICAL TRIAL: NCT03626194
Title: Prospective Evaluation of the Efficacy and Safety of Endoscopic Tissue Apposition
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 16-1826
Record Dates: First submitted 2018-08-02; First posted 2018-08-10 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Endoscopic Tissue Apposition; Endoscopic Suturing; Endoscopic Clipping; Bariatric Endoscopy; Transoral Outlet Reduction; Endoscopic Sleeve Gastroplasty

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a prospective registry of patients undergoing endoscopic suturing and/or clip placement at our institution to assess the efficacy and safety of endoscopic tissue apposition.

1.1 Hypothesis: Endoscopic tissue apposition is efficacious and safe in the practice of gastrointestinal endoscopy.

1.2 Aims: To prospectively evaluate the efficacy and safety of Endoscopic Tissue Apposition in the practice of gastrointestinal endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patients>18 years of age undergoing endoscopy for any of the following indications:

Indications for Tissue Apposition:

* Closure of perforations
* Closure of full thickness defects created during endoscopic full thickness resection
* Closure of defects after endoscopic submucosal dissection and endoscopic mucosal resection
* Closure of mucosotomy after Peroral Endoscopic Myotomy (POEM)
* Stent fixation
* Closure of fistulas
* Natural Orifice Transluminal Endoscopic Surgery defect closures
* Post-bariatric surgery gastrojejunal anastomosis and gastric pouch revision (transoral outlet repair)
* Primary endoscopic sleeve gastroplasty

Exclusion Criteria:

* Patients unable or unwilling to provide consent
* Pregnant patients
* Coagulation disorders (INR >1.8, platelet <50,000)
* GI Bleeding
* Hemodynamic instability
* Enrollment in another device or drug study that may confound the results

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A prospective database/registry of patients undergoing endoscopic tissue apposition will be formed. Women and minorities will be included as they are frequently found to have indications for which endoscopic tissue apposition may be indicated.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-12-12 (Actual); Primary Completion 2025-12-16 (Estimated); Study Completion 2026-12-16 (Estimated)

PRIMARY OUTCOMES:
Technical and clinical success in endoscopic tissue apposition | From baseline to one year
  Successful completion of endoscopic suturing/clipping and measured as clinical symptom improvement as well as objective evidence of resolution / improvement of underlying pathology / confirmed with radiologic contrast studies as needed..
Adverse Events | From baseline to one year
  Based on ASGE criteria

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States